CLINICAL TRIAL: NCT02672748
Title: Growing Resilience: an RCT on the Health Impact of Gardens With Wind River Indian Reservation
Brief Title: Growing Resilience in Wind River Indian Reservation
Acronym: GR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wyoming (Other)
Collaborators: Blue Mountain Associates, Incorporated (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Eastern Shoshone Tribal Health (Unknown); Action Resources International (Other); National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH); Wind River Development Fund (WRDF) (Unknown)
Responsible Party: Principal Investigator, Christine Porter, Associate Professor, University of Wyoming
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL126666-01A1 (NIH); R01HL126666-01A1 (NIH)
Record Dates: First submitted 2015-11-09; First posted 2016-02-03 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Obesity; Overweight; Diabetes
Keywords: garden; Native American; BMI; Emotional health; Physical health
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus; Psychological Well-Being | interventions — Gardens

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary data analyst will not know which set of results are from people in the gardening vs. the control condition.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gardening (Experimental): Receiving two years of technical, labor and financial support in starting, growing, and harvesting from a home food garden.
  Interventions: Other: Garden
- Control (No Intervention): The control families receive a garden as a delayed intervention after two years.

INTERVENTIONS:
Other: Garden — Two years of financial and technical home gardening support for new gardeners
  Arms: Gardening

SUMMARY:
The Growing Resilience research leverages reservation-based assets of land, family, culture, and front-line tribal health organizations to develop and evaluate home food gardens as a family-based health promotion intervention to reduce disparities suffered by Native Americans in nearly every measure of health. Home gardening interventions show great promise for enabling families to improve their health, and this study aims to fulfill that promise with university and Wind River Indian Reservation partners. The investigators will develop an empowering, scalable, and sustainable family-based health promotion intervention with, by, and for Native American families and conduct the first RCT to assess the health impacts of home gardens.

DETAILED DESCRIPTION:
The intervention is comprised of designing and providing two years of support for home gardens. Families randomized to intervention will receive the following supports and services:

1. Blue Mountain Associates will host a gardening workshop to include crop planning, receipt of customized guides to the crops the family selects (these are currently in development and will be ready by 2015), and hands-on basic skills training (mid-April). CHRs and interested local healthcare providers will also participate in workshops to help them prepare for supporting gardeners.
2. BMA's garden manager and assistant(s) will visit each family to help the family install a garden and will provide the family with all needed supplies (late April to early May). Based on garden harvest measures collected in the Food Dignity project and the large gardens preferred by families in the pilot, the minimum garden size will be 80 sq. ft. with at least 30 sq. ft. devoted to crops other than corn and potatoes. The manager will design at least part of each garden in a way that allows the least physically able family members to participate in gardening.
3. BMA will host a Facebook support and networking group for gardeners, with ARI, BMA, and UW gardening experts providing advice as needed.
4. BMA's staff will visit each gardening family at least twice more during the growing season and will be available throughout the season for phone consultations and Facebook advice. For all years, the BMA garden manager will track actual intervention support provided to each family (e.g., timing and number of visits, training and supplies provided).

The University of Wyoming research team will collect health measures before and at the end of each gardening season with gardening and control families for two years, after which the control families also receive the gardening intervention. The investigators anticipate enrolling about 100 families into the study with 400 (half adults, half children) people participating in the health measures.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as having one or more household members who are enrolled in a tribe
* express interest in having a food garden
* express willingness to wait to create a food garden for two years if randomized to control
* live within the boundaries of Wind River Indian Reservation, including the City of Riverton.
* if the household has two or more adults, that at least two adults in the household express willingness to participate in the semi-annual data gathering for two years.

Exclusion Criteria:

* had a home food garden plot in the previous year that is over 30 square feet in area.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Adult BMI change | Change from baseline at 2 years
  With four data points, every 6 months. Researcher-measured height (stadiometer) and Tanita body composition scale.

SECONDARY OUTCOMES:
Mental Health change | Change from baseline at 2 years
  measured by SF12 survey
Physical Health change | Change from baseline at 2 years
  measured by SF12 survey
Food security change | Change from baseline at 2 years
  measured by sub-set of USDA survey
Self-efficacy in gardening change | Change from baseline at 2 years
  by survey
Pain change | Change from baseline at 2 years
  by survey
Blood pressure change | Change from baseline at 2 years
  researcher-measured with bp monitor
hand strength change | Change from baseline at 2 years
  researcher-measured with dynamometer
waist circumference change | Change from baseline at 2 years
  researcher-measured with spring-loaded tape measure
beta-carotene change | Change from baseline at 2 years
  whole blood draw and assay
Hb A1C change | Change from baseline at 2 years
  whole blood draw and assay
cholesterol change | Change from baseline at 2 years
  whole blood draw and assay
triglycerides change | Change from baseline at 2 years
  whole blood draw and assay
vitamin D change | Change from baseline at 2 years
  whole blood draw and assay
child BMI z-score change | Change from baseline at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Porter, PhD, Principal Investigator — University of Wyoming
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be made available to each individual participant, but otherwise only the data summaries will be made available to non-partner parties unless individually arranged and approved by the IRB and project Community Advisory Board. The Northern Arapaho and the Eastern Shoshone tribes co-own the data with the research teams (and Eastern Shoshone Tribal Health and Northern Arapaho Tribal Health are entities of the tribal governments).

REFERENCES:
- [Derived] Naschold F, Porter CM. BMI Status and Trends among Native American Family Members Participating in the Growing Resilience Home Garden Study. Curr Dev Nutr. 2022 Jun 3;6(7):nzac100. doi: 10.1093/cdn/nzac100. eCollection 2022 Jul. PMID 35898313
- [Derived] Porter CM, Wechsler AM, Hime SJ, Naschold F. Adult Health Status Among Native American Families Participating in the Growing Resilience Home Garden Study. Prev Chronic Dis. 2019 Aug 22;16:E113. doi: 10.5888/pcd16.190021. PMID 31441769
- [Derived] Porter CM, Wechsler AM, Naschold F, Hime SJ, Fox L. Assessing health impacts of home food gardens with Wind River Indian Reservation families: protocol for a randomised controlled trial. BMJ Open. 2019 Apr 3;9(4):e022731. doi: 10.1136/bmjopen-2018-022731. PMID 30948560
- See also: website for the project — http://www.growingresilience.org